CLINICAL TRIAL: NCT03016117
Title: Anesthetic Efficacy of PECS II Block and Parasternal Block for Quadrantectomy With or Without Axillary Dissection
Brief Title: Anesthetic Efficacy of PECS II Block and Parasternal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Emiliano Petrucci, MD, San Salvatore Hospital of L'Aquila
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SanSalvatoreH
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pecs II block and parasternal block (Experimental): Pecs II block and parasternal block performed to provide anesthesia of breast, before of quadrantectomy with or without axillary dissection. Pecs II block performed at the 4th rib level and 20 ml of 0.5% Levobupivacaine injected, and parasternal block performed at the level of the 2nd and 4th intercostal space level, and 4 ml of 0.375% Levobupivacaine injected
  Interventions: Procedure: Pecs II block and parasternal block

INTERVENTIONS:
Procedure: Pecs II block and parasternal block — The Pecs II block will be performed under ultrasound guidance, at fourth rib level, on the axillary line, into the fascial plane between pectoralis minor muscle and serratus muscle. The parasternal block will be performed under ultrasound guidance, at the second and fourth intercostal space, between the pectoralis major muscle and the intercostal muscles, near to the external intercostal membrane.

SUMMARY:
The study evaluate the anesthetic efficacy of Pecs II block II and parasternal block during quadrantectomy with or without axillary dissection, in breast cancer surgery

DETAILED DESCRIPTION:
All patients receive Pecs II block and parasternal block, under ultrasound guidance. Pecs II block, performed at the 4th rib level, and parasternal block performed at the level of the 2nd and 4th intercostal space level. Data on the anesthesia, side effects and pain, will be recorded

ELIGIBILITY:
Inclusion Criteria:

* patients who need of quadrantectomy with or without axillary dissection
* ASA I-III patients
* age between 18 and 75 years
* filled informed consent

Exclusion Criteria:

* pregnant women
* obesity (BMI > 39,99)
* radical mastectomy
* ASA IV patients
* chest wall abnormalities
* neurological disorders
* septic status
* chest skin infections
* coagulopathies

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Anesthetic efficacy | The anesthetic efficacy was assessed in the first 72 hours, after block
  The anesthetic efficacy is tested by cold and touch test

SECONDARY OUTCOMES:
Painkillers request | The painkillers request was assessed in the first 72 hours, after surgery
  mg of morphine
Side effects | The side effects recorded in the first 72 hours, after surgery
  Nausea, vomiting, local anesthetic systemic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Pierfrancesco Fusco, MDD, Principal Investigator — San Salvatore Academic Hospital
Locations (1):
- San Salvatore Academic Hospital, Coppito, L'Aquila, Italy

IPD SHARING:
Plan to Share IPD: No